CLINICAL TRIAL: NCT04606745
Title: Increase of Handgrip Strength After the Use of Removable Partial Dentures.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Gerardo F Fasce Pineda, MD, MD, University of Chile
Other Study IDs: HDEN
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sarcopenia
Keywords: removable partial dentures
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A common goal of the health professions is to keep the elderly functional, preventing sarcopenia and frailty. Is there an association between handgrip strength in partially edentulous elderlies after completing their dentition with removable partial dentures?

DETAILED DESCRIPTION:
A common goal of the health professions is to keep the elderly functional, preventing sarcopenia and frailty. Is there an association between handgrip strength in partially edentulous elderlies after completing their dentition with removable partial dentures?

ELIGIBILITY:
Inclusion Criteria:

* agree to participate by signing the voluntary informed consent form
* qualify according to the Eichner Index in any of the categories that represent the loss of premolars and molars: B3-B4-C1-and C2.

Exclusion Criteria:

* not accepting to participate
* cognitive or auditory sensory impairment-
* being dependent in activities of daily living
* belonging to another category of the Eichner Index

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Independent octogenarians that consulted in centers of the greater metropolitan area of Santiago, Chile, in search of solving their lack of posterior teeth with dental prostheses
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | 18 months
  role of use of removable partial dentures (RPD) in handgrip strength in octogenarians

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Chile, Santiago, Chile